CLINICAL TRIAL: NCT07330869
Title: Effects of Warfarin Therapy on Semen Quality, DNA Integrity, Hormonal Profile and Molecular Alterations in Male Patients Undergoing Cardiac Surgery: A Prospective Comparative Pilot Study
Brief Title: Warfarin Effects on Male Fertility After Cardiac Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: Città di Lecce Hospital, GVM Care & Research (Other)
Responsible Party: Sponsor
Other Study IDs: WARF-SEMIN-2025-01
Record Dates: First submitted 2025-12-15; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Male Infertility; Heart Valve Disease
Keywords: warfarin; male infertility; Semen quality; Sperm DNA fragmentation; Mitochondrial function; Inflammation; Mechanical heart valve; Cardiac surgery; Oral anticoagulation; Vitamin K antagonists; Reproductive hormones; anticoagulation
MeSH Terms: conditions — Infertility, Male; Heart Valve Diseases; Inflammation | interventions — Semen Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Semen samples and blood samples will be collected and retained for planned analyses, including standard semen parameters, sperm DNA fragmentation assessment, hormonal assays and exploratory molecular analyses related to mitochondrial function, oxidative stress, inflammatory markers, and protein expression.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Long-term Warfarin Group: Male patients undergoing cardiac surgery with an indication for lifelong oral anticoagulation with warfarin, typically after mechanical heart valve replacement. Warfarin therapy is prescribed as part of standard clinical care and is not assigned by the study.
  Interventions: Other: Semen analysis, sperm DNA fragmentation and hormonal evaluation
- Short-term Warfarin Group: Male patients undergoing cardiac surgery with an indication for short-term postoperative warfarin therapy (approximately three months), such as after valve repair or bioprosthetic valve implantation. Anticoagulation is administered according to standard clinical practice and not determined by the study protocol.
  Interventions: Other: Semen analysis, sperm DNA fragmentation and hormonal evaluation
- Control Group (No Long-term Anticoagulation): Male patients undergoing cardiac surgery without an indication for long-term oral anticoagulation beyond routine perioperative prophylaxis. These patients serve as a comparison group and do not receive chronic warfarin therapy.
  Interventions: Other: Semen analysis, sperm DNA fragmentation and hormonal evaluation

INTERVENTIONS:
Other: Semen analysis, sperm DNA fragmentation and hormonal evaluation — Participants undergo standardized study assessments including semen analysis according to WHO criteria, sperm DNA fragmentation assessment, hormonal blood tests, andrological ultrasound, and exploratory molecular analyses of spermatozoa (mitochondrial function, oxidative stress markers, inflammatory mediators, and protein expression). All assessments are performed for observational and research purposes only and do not guide or modify clinical treatment.

SUMMARY:
Young male patients undergoing cardiac surgery may require oral anticoagulation with warfarin either lifelong, such as after mechanical valve replacement, or for a limited postoperative period, for example following valve repair or bioprosthetic valve implantation. Although the teratogenic effects of warfarin during pregnancy are well established, prospective clinical data on the potential impact of warfarin therapy on male reproductive health are scarce. This gap is particularly relevant for patients of reproductive age who may have a present or future desire for fatherhood.

Warfarin acts as a vitamin K antagonist by inhibiting the vitamin K epoxide reductase complex, thereby reducing the availability of functional vitamin K. Beyond its role in coagulation, vitamin K is increasingly recognized as an important regulator of spermatogenesis, mitochondrial function, oxidative balance, and steroid hormone synthesis. Experimental and translational evidence suggests that disruption of vitamin K-dependent pathways may impair sperm quality, DNA integrity, mitochondrial bioenergetics, and reproductive hormone homeostasis. In addition, warfarin exposure has been associated with increased oxidative stress and inflammatory responses, both of which are known contributors to male infertility.

Despite these biologically plausible mechanisms, no prospective observational studies have systematically evaluated semen parameters, sperm DNA fragmentation, hormonal profiles, inflammatory markers, and advanced molecular sperm alterations in men exposed to warfarin after cardiac surgery. Consequently, structured andrological assessment is rarely incorporated into routine preoperative counseling or postoperative follow-up in this population.

This prospective pilot observational study aims to investigate the association between warfarin therapy and male reproductive health in patients undergoing elective cardiac surgery. Male patients aged 18 to 50 years will be enrolled and observed in three cohorts based on clinical indication for anticoagulation: (1) long-term warfarin therapy following mechanical valve replacement; (2) short-term warfarin therapy (approximately three months) after selected cardiac procedures; and (3) a control cohort undergoing cardiac surgery without an indication for long-term oral anticoagulation beyond standard perioperative prophylaxis.

Participants will undergo comprehensive andrological assessments at baseline and during follow-up up to 12 months after surgery. Evaluations will include semen analysis according to World Health Organization guidelines, assessment of sperm DNA fragmentation, reproductive hormonal profiles, and seminal inflammatory markers. Exploratory analyses will assess mitochondrial function, oxidative stress, and molecular alterations in spermatozoa. Detailed warfarin exposure data, including dose, cumulative exposure, international normalized ratio values, and time in therapeutic range, will be collected to explore potential exposure-response relationships.

As a pilot study, the primary aims are to assess feasibility and generate preliminary clinical evidence to inform future larger studies. The findings may contribute to improved clinical counseling, fertility preservation strategies, and integration of reproductive health considerations into the multidisciplinary management of young male cardiac surgery patients.

DETAILED DESCRIPTION:
This prospective, comparative, pilot observational study is designed to investigate the effects of warfarin therapy on male reproductive health in patients undergoing elective cardiac surgery, integrating conventional andrological assessment with inflammatory, hormonal, and exploratory molecular analyses.

Young male patients undergoing cardiac surgery may require oral anticoagulation with warfarin either lifelong, most commonly after mechanical heart valve replacement, or for a limited postoperative period following selected procedures such as valve repair or bioprosthetic valve implantation. Although the teratogenic effects of warfarin during pregnancy are well established, prospective clinical data addressing its potential impact on male reproductive health are scarce. This knowledge gap is particularly relevant for patients of reproductive age who may have a present or future desire for fatherhood and for whom fertility-related counseling is increasingly important.

Warfarin exerts its anticoagulant effect through inhibition of the vitamin K epoxide reductase (VKOR) complex, resulting in reduced availability of biologically active vitamin K. Beyond its role in coagulation, vitamin K-dependent pathways are involved in key aspects of male reproductive physiology, including spermatogenesis, mitochondrial bioenergetics, oxidative stress regulation, inflammatory signaling, and steroid hormone synthesis. Experimental and translational evidence suggests that disruption of these pathways may impair semen quality, sperm DNA integrity, mitochondrial function, and endocrine homeostasis, while promoting oxidative stress and inflammatory responses known to contribute to male infertility. However, these mechanisms have not been systematically explored in prospective clinical studies involving men exposed to warfarin after cardiac surgery.

The study adopts a prospective cohort design with a comparative approach and includes three groups of male patients stratified according to clinical indication for anticoagulation: (1) patients receiving long-term warfarin therapy following mechanical valve replacement; (2) patients receiving short-term postoperative warfarin therapy, typically for approximately three months, after selected cardiac surgical procedures; and (3) a control group undergoing cardiac surgery without indication for long-term oral anticoagulation beyond standard perioperative prophylaxis. This design allows evaluation of different exposure patterns, including chronic exposure, transient exposure, and non-exposure, and supports exploratory assessment of exposure-response relationships and reversibility after treatment discontinuation.

Participants undergo structured and standardized andrological evaluations at baseline (preoperative) and during longitudinal follow-up up to 12 months after surgery. Conventional semen analysis is performed according to World Health Organization (WHO) guidelines and includes assessment of sperm concentration, progressive motility, morphology, and related semen parameters. Sperm DNA integrity is evaluated through measurement of the sperm DNA fragmentation index (DFI) using the sperm chromatin dispersion (SCD) assay.

Reproductive endocrine function is assessed through serial measurement of serum reproductive hormones, including follicle-stimulating hormone (FSH), luteinizing hormone (LH), total testosterone, sex hormone-binding globulin (SHBG), prolactin, and thyroid-stimulating hormone (TSH), using standardized laboratory immunoassay methods.

Local inflammatory processes within the male reproductive tract are investigated through assessment of seminal inflammatory mediators, including interleukin-6 (IL-6), tumor necrosis factor-alpha (TNF-α), prostaglandin E2 (PGE2), and prostaglandin F2α (PGF2α). These biomarkers are measured using standardized enzyme-linked immunosorbent assay (ELISA) techniques and evaluated in relation to semen quality parameters.

To provide mechanistic insight beyond conventional clinical and laboratory assessments, exploratory molecular analyses are performed on spermatozoa. These analyses include evaluation of mitochondrial function and bioenergetics, assessment of oxidative stress-related parameters, and analysis of selected proteins involved in sperm energy metabolism and motility, using validated laboratory techniques. These exploratory investigations are intended to characterize molecular alterations potentially associated with warfarin exposure and to generate hypotheses for future mechanistic studies.

Detailed warfarin exposure data are collected prospectively from clinical records and anticoagulation monitoring systems, including daily and cumulative dosing information, international normalized ratio (INR) measurements, and quality of anticoagulation control over time as reflected by time in therapeutic range (TTR). These exposure variables are used to support exploratory correlation analyses with reproductive, inflammatory, and molecular outcomes, as well as evaluation of potential reversibility of observed alterations in patients receiving short-term warfarin therapy after treatment discontinuation.

Sexual and reproductive function is further characterized through validated questionnaires assessing sexual function, including the International Index of Erectile Function-5 (IIEF-5), and through collection of exploratory reproductive outcomes, such as desire for paternity and occurrence of partner pregnancies during follow-up.

As a pilot study, the primary objectives are to assess feasibility, characterize longitudinal changes in male reproductive parameters, and generate preliminary clinical and mechanistic data to inform the design of future larger-scale studies. The findings are expected to contribute to improved fertility-related counseling, consideration of fertility preservation strategies, and integration of reproductive health assessment into the multidisciplinary management of young male patients undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male sex, age between 18 and 50 years;
* Scheduled for elective cardiac surgery (valve replacement, valve repair, or other cardiac procedures) with or without indication to Warfarin therapy;
* Ability and willingness to provide semen samples at scheduled timepoints;
* No previous diagnosis of male infertility documented in medical records;
* Signed informed consent.

Exclusion Criteria:

* Known severe testicular pathology (for example, untreated high-grade varicocele, history of cryptorchidism, orchiectomy, testicular tumors);
* Prior chemotherapy or pelvic radiotherapy;
* Current or recent use of anabolic steroids or other drugs known to strongly impair spermatogenesis;
* Known endocrine disorders affecting spermatogenesis (for example, untreated hypogonadism, hyperprolactinaemia, severe thyroid disease);
* Active genitourinary infection at the time of evaluation;
* Life expectancy less than 12 months or clinical conditions preventing adherence to follow-up.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study will enroll male patients aged 18 to 50 years undergoing elective cardiac surgery at a high-volume cardiac surgery center. Participants will include individuals requiring either lifelong Warfarin therapy (mechanical heart valve replacement), short-term postoperative Warfarin therapy (e.g., mitral valve repair or bioprosthetic valve implantation), or no long-term anticoagulation beyond routine perioperative prophylaxis.
  Eligible patients must have no previous diagnosis of male infertility, must be able and willing to provide semen samples at scheduled follow-up timepoints, and must provide written informed consent. Patients with severe testicular disease, prior chemotherapy or radiotherapy, endocrine disorders affecting spermatogenesis, active genitourinary infection, or current/recent use of anabolic steroids or medications known to impair spermatogenesis will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Change in sperm concentration over time | Baseline (T0) to 6 months (T2) and 12 months (T3)
  Change in sperm concentration expressed as millions of spermatozoa per milliliter (millions/mL), assessed by standard semen analysis performed according to World Health Organization (WHO) guidelines. Correlation between warfarin exposure status (long-term exposure, short-term exposure, or no exposure) and changes in sperm concentration over time will be evaluated.
Change in progressive sperm motility over time | Baseline (T0) to 6 months (T2) and 12 months (T3)
  Change in progressive sperm motility expressed as percentage (%), assessed by standard semen analysis according to World Health Organization (WHO) guidelines. Correlation between warfarin exposure status (long-term exposure, short-term exposure, or no exposure) and changes in progressive sperm motility over time will be evaluated.
Change in sperm morphology over time | Baseline (T0) to 6 months (T2) and 12 months (T3)
  Change in the percentage (%) of spermatozoa with normal morphology, assessed using strict criteria as part of standard semen analysis according to World Health Organization (WHO) guidelines. Correlation between warfarin exposure status (long-term exposure, short-term exposure, or no exposure) and changes in sperm morphology over time will be evaluated.

SECONDARY OUTCOMES:
Change in sperm DNA fragmentation index (DFI) | Baseline (T0), 3 months (T1), 6 months (T2), and 12 months (T3)
  Change in sperm DNA fragmentation index (DFI), assessed using a validated assay (sperm chromatin dispersion method), between baseline and follow-up timepoints in warfarin-exposed and control groups.
Change in serum follicle-stimulating hormone (FSH) levels | Baseline (T0), 3 months (T1), 6 months (T2), and 12 months (T3)
  Change in serum follicle-stimulating hormone (FSH) levels, measured in international units per liter (IU/L) using standard immunoassay methods, evaluated over time and compared between study groups.
Change in serum luteinizing hormone (LH) levels | Baseline (T0), 3 months (T1), 6 months (T2), and 12 months (T3)
  Change in serum luteinizing hormone (LH) levels, measured in international units per liter (IU/L) using standard immunoassay methods, evaluated over time and compared between study groups.
Change in serum total testosterone levels | Baseline (T0), 3 months (T1), 6 months (T2), and 12 months (T3)
  Change in serum total testosterone levels, measured in nanograms per deciliter (ng/dL) using standard immunoassay methods, evaluated over time and compared between study groups.
Change in serum sex hormone-binding globulin (SHBG) levels | Baseline (T0), 3 months (T1), 6 months (T2), and 12 months (T3)
  Change in serum sex hormone-binding globulin (SHBG) levels, measured in nanomoles per liter (nmol/L) using standard immunoassay methods, evaluated over time and compared between study groups.
Change in serum prolactin levels | Baseline (T0), 3 months (T1), 6 months (T2), and 12 months (T3)
  Change in serum prolactin levels, measured in nanograms per milliliter (ng/mL) using standard immunoassay methods, evaluated over time and compared between study groups.
Change in serum thyroid-stimulating hormone (TSH) levels | Baseline (T0), 3 months (T1), 6 months (T2), and 12 months (T3)
  Change in serum thyroid-stimulating hormone (TSH) levels, measured in milli-international units per liter (mIU/L) using standard immunoassay methods, evaluated over time and compared between study groups.
Correlation between mean daily warfarin dose and changes in semen parameters | Baseline (T0), 3 months (T1), 6 months (T2), and 12 months (T3)
  Correlation between mean daily warfarin dose, expressed in milligrams per day (mg/day), and changes from baseline in semen parameters assessed by standard semen analysis according to World Health Organization (WHO) guidelines, in warfarin-exposed patients.
Correlation between cumulative warfarin dose and changes in semen parameters | Baseline (T0), 3 months (T1), 6 months (T2), and 12 months (T3)
  Correlation between cumulative warfarin dose, expressed in milligrams (mg), and changes from baseline in semen parameters assessed by standard semen analysis according to World Health Organization (WHO) guidelines, in warfarin-exposed patients.
Correlation between time in therapeutic range and changes in semen parameters | Baseline (T0), 3 months (T1), 6 months (T2), and 12 months (T3)
  Correlation between time in therapeutic range (TTR), expressed as percentage (%), and changes from baseline in semen parameters assessed by standard semen analysis according to World Health Organization (WHO) guidelines, in warfarin-exposed patients.
Correlation between warfarin exposure and changes in sperm DNA fragmentation index | Baseline (T0), 3 months (T1), 6 months (T2), and 12 months (T3)
  Correlation between warfarin exposure variables (mean daily dose [mg/day], cumulative dose [mg], and time in therapeutic range [%]) and changes from baseline in sperm DNA fragmentation index (DFI), expressed as percentage (%), assessed using the sperm chromatin dispersion (SCD) assay.
Reversibility of changes in semen parameters after short-term warfarin discontinuation | From 3 to 6 months after surgery (T1 to T2)
  Evaluation of reversibility of changes from baseline in semen parameters assessed by standard semen analysis according to World Health Organization (WHO) guidelines, between 3 and 6 months after surgery (T1 to T2), in patients receiving short-term warfarin therapy.
Reversibility of changes in sperm DNA fragmentation index after short-term warfarin discontinuation | From 3 months (T1) to 6 months (T2) after surgery
  Evaluation of reversibility of changes from baseline in sperm DNA fragmentation index (DFI), expressed as percentage (%), assessed using the sperm chromatin dispersion (SCD) assay, between 3 and 6 months after surgery (T1 to T2), in patients receiving short-term warfarin therapy.
Correlation between seminal interleukin-6 (IL-6) levels and semen parameters | Baseline (T0), 3 months (T1), 6 months (T2), and 12 months (T3)
  Correlation between seminal interleukin-6 (IL-6) concentration, measured using a standardized enzyme-linked immunosorbent assay (ELISA), and changes from baseline in semen parameters assessed by standard semen analysis according to World Health Organization (WHO) guidelines.
Correlation between seminal tumor necrosis factor-alpha (TNF-α) levels and semen parameters | Baseline (T0), 3 months (T1), 6 months (T2), and 12 months (T3)
  Correlation between seminal tumor necrosis factor-alpha (TNF-α) concentration, measured using a standardized enzyme-linked immunosorbent assay (ELISA), and changes from baseline in semen parameters assessed by standard semen analysis according to World Health Organization (WHO) guidelines.
Correlation between seminal prostaglandin E2 (PGE2) levels and semen parameters | Baseline (T0), 3 months (T1), 6 months (T2), and 12 months (T3)
  Correlation between seminal prostaglandin E2 (PGE2) concentration, measured using a standardized enzyme-linked immunosorbent assay (ELISA), and changes from baseline in semen parameters assessed by standard semen analysis according to World Health Organization (WHO) guidelines.
Correlation between seminal prostaglandin F2α (PGF2α) levels and semen parameters | Baseline (T0), 3 months (T1), 6 months (T2), and 12 months (T3)
  Correlation between seminal prostaglandin F2α (PGF2α) concentration, measured using a standardized enzyme-linked immunosorbent assay (ELISA), and changes from baseline in semen parameters assessed by standard semen analysis according to World Health Organization (WHO) guidelines.
Exploratory assessment of mitochondrial function in spermatozoa | Baseline (T0), 3 months (T1), 6 months (T2), and 12 months (T3)
  Exploratory evaluation of mitochondrial function in spermatozoa, assessed using validated bioenergetic assays evaluating mitochondrial respiratory activity and related functional parameters.
Exploratory assessment of oxidative stress markers in spermatozoa | Baseline (T0), 3 months (T1), 6 months (T2), and 12 months (T3)
  Exploratory evaluation of oxidative stress-related parameters in spermatozoa, assessed using validated assays measuring reactive oxygen species production and lipid peroxidation markers.
Exploratory assessment of sperm protein expression involved in bioenergetics and motility | Baseline (T0), 3 months (T1), 6 months (T2), and 12 months (T3)
  Exploratory evaluation of the expression of selected sperm proteins involved in bioenergetics and motility, assessed using validated protein analysis techniques.
Change in sexual function assessed by the International Index of Erectile Function-5 (IIEF-5) | Baseline (T0), 3 months (T1), 6 months (T2), and 12 months (T3)
  Change in sexual function assessed using the International Index of Erectile Function-5 (IIEF-5) questionnaire, expressed as total score on a validated scale, evaluated over time and compared between study groups.
Desire for paternity over time | Baseline (T0), 3 months (T1), 6 months (T2), and 12 months (T3)
  Assessment of desire for paternity, recorded as a categorical variable (presence or absence of desire for fatherhood), evaluated over time and compared between study groups.
Occurrence of partner pregnancies during follow-up | Baseline (T0), 3 months (T1), 6 months (T2), and 12 months (T3)
  Occurrence of partner pregnancies during the follow-up period, assessed as incidence of pregnancies reported by participants and compared between study groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Città di Lecce Hospital - Department of Cardiac Surgery, Lecce, LE, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Popov A, Belij S, Subota V, Zolotarevski L, Mirkov I, Kataranovski D, Kataranovski M. Oral warfarin affects peripheral blood leukocyte IL-6 and TNFalpha production in rats. J Immunotoxicol. 2013 Jan-Mar;10(1):17-24. doi: 10.3109/1547691X.2012.684159. Epub 2012 Jul 13. PMID 22793260
- [Result] Azenabor A, Ekun AO, Akinloye O. Impact of Inflammation on Male Reproductive Tract. J Reprod Infertil. 2015 Jul-Sep;16(3):123-9. PMID 26913230
- [Result] Ma H, Zhang BL, Liu BY, Shi S, Gao DY, Zhang TC, Shi HJ, Li Z, Shum WW. Vitamin K2-Dependent GGCX and MGP Are Required for Homeostatic Calcium Regulation of Sperm Maturation. iScience. 2019 Apr 26;14:210-225. doi: 10.1016/j.isci.2019.03.030. Epub 2019 Mar 29. PMID 30981116
- [Result] Shiba S, Ikeda K, Horie-Inoue K, Azuma K, Hasegawa T, Amizuka N, Tanaka T, Takeiwa T, Shibata Y, Koji T, Inoue S. Vitamin K-Dependent gamma-Glutamyl Carboxylase in Sertoli Cells Is Essential for Male Fertility in Mice. Mol Cell Biol. 2021 Mar 24;41(4):e00404-20. doi: 10.1128/MCB.00404-20. Print 2021 Mar 24. PMID 33526452
- [Result] Alfano M, Pederzoli F, Locatelli I, Ippolito S, Longhi E, Zerbi P, Ferrari M, Brendolan A, Montorsi F, Drago D, Andolfo A, Nebuloni M, Salonia A. Impaired testicular signaling of vitamin A and vitamin K contributes to the aberrant composition of the extracellular matrix in idiopathic germ cell aplasia. Fertil Steril. 2019 Apr;111(4):687-698. doi: 10.1016/j.fertnstert.2018.12.002. PMID 30929729
- [Result] Shirakawa H, Ohsaki Y, Minegishi Y, Takumi N, Ohinata K, Furukawa Y, Mizutani T, Komai M. Vitamin K deficiency reduces testosterone production in the testis through down-regulation of the Cyp11a a cholesterol side chain cleavage enzyme in rats. Biochim Biophys Acta. 2006 Oct;1760(10):1482-8. doi: 10.1016/j.bbagen.2006.05.008. Epub 2006 Jun 6. PMID 16844298
- [Result] Sanyaolu AO, Oremosu AA, Osinubi AA, Vermeer C, Daramola AO. Warfarin-induced vitamin K deficiency affects spermatogenesis in Sprague-Dawley rats. Andrologia. 2019 Nov;51(10):e13416. doi: 10.1111/and.13416. Epub 2019 Oct 1. PMID 31576592
- [Result] Regitz-Zagrosek V, Roos-Hesselink JW, Bauersachs J, Blomstrom-Lundqvist C, Cifkova R, De Bonis M, Iung B, Johnson MR, Kintscher U, Kranke P, Lang IM, Morais J, Pieper PG, Presbitero P, Price S, Rosano GMC, Seeland U, Simoncini T, Swan L, Warnes CA; ESC Scientific Document Group. 2018 ESC Guidelines for the management of cardiovascular diseases during pregnancy. Eur Heart J. 2018 Sep 7;39(34):3165-3241. doi: 10.1093/eurheartj/ehy340. No abstract available. PMID 30165544
- [Result] Chan WS, Anand S, Ginsberg JS. Anticoagulation of pregnant women with mechanical heart valves: a systematic review of the literature. Arch Intern Med. 2000 Jan 24;160(2):191-6. doi: 10.1001/archinte.160.2.191. PMID 10647757
- [Result] Hall JG, Pauli RM, Wilson KM. Maternal and fetal sequelae of anticoagulation during pregnancy. Am J Med. 1980 Jan;68(1):122-40. doi: 10.1016/0002-9343(80)90181-3. PMID 6985765